CLINICAL TRIAL: NCT07189377
Title: Lung Transplantation Using Hepatitis B Positive Donors to Hepatitis B Negative Recipients Using Ex-Vivo Treatment of Organs: A Safety Trial
Brief Title: Combined Light, ExVivo, and Antivirals for Recipients of Lungs From HBV Donors
Acronym: CLEAR-HBV
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-6051
Record Dates: First submitted 2025-09-09; First posted 2025-09-23 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Hepatitis B Virus (HBV); Lung Transplant Recipient
Keywords: HBV Disease; EVLP; lung transplant
MeSH Terms: conditions — Hepatitis B | interventions — entecavir; hepatitis B hyperimmune globulin

STUDY DESIGN:
Intervention Model Description: The antiviral used are both approved drugs (entecavir and HBIG) but being used for a new indication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UV Light + Short-course Entecavir/HBIG (Experimental): Patients will receive lungs from HBV NAT+ donors, which will be treated with UV light therapy during ex-vivo perfusion. Patients will also receive Entecavir and HBIG prophylaxis in the immediate peri-operative period.
  Interventions: Drug: Entecavir; Biological: HBIG; Device: EVLP UV Light Treatment

INTERVENTIONS:
Drug: Entecavir — Recipients will receive 1mg administered orally, beginning pre-transplant as soon as the patient arrives to the hospital for surgery, and then 1mg post-operatively administered orally or via nasogastric tube once daily for 28 days.
Biological: HBIG — Recipients will receive 4500 IU intravenously pre-transplant and then at day 3 and 7 post-transplant (3 doses total).
Device: EVLP UV Light Treatment — UV light therapy will be administered to the organ during EVLP prior to transplantation. For minimum 2 hours, maximum 6 hours (duration determined by time clinically required for EVLP based on standard clinical assessment of lung).

SUMMARY:
The aim of the study is to show that transplantation of lungs from Hepatitis B-infected donors is safe when using EVLP with UV light inactivation plus antivirals

DETAILED DESCRIPTION:
The success of transplantation is significantly hindered by the lack of sufficient available donors. Many potential donor organs are not fully utilized in clinical transplantation because donors have chronic viral infections. Currently, donors with chronic hepatitis B virus (HBV) infection are utilized by typically providing nucleoside analogues such as entecavir or lamivudine plus/minus several doses of HBIG. The entecavir or lamivudine are typically given either life-long in liver transplants or for 1 year in non-liver transplants. Donors with chronic HBV infection are Core Antibody positive (HBcAb +ve). These donors carry chronic virus but may be NAT positive or NAT negative. HBcAb+ve donors are routinely used, but NAT positive donors are typically not used. The Toronto lung transplant program commonly applies Ex Vivo Lung Perfusion (EVLP) to organs. This allows for treatment of organs prior to transplantation. The investigators have shown that UV light administered on the EVLP circuit can substantially decrease the amount of infectious virus. Such a strategy was previously employed with hepatitis C virus. The aim of the study is to show that transplantation of organs from HBV NAT+ve donors is safe with the use of UV light treatment on EVLP combined with post-transplant antivirals for the recipient (HBIG and entecavir). The investigators hypothesize that rates of HBV transmission to recipients will be prevented by the use of this approach and any HBV transmission that does occur will be readily treatable. This will be a small pilot study to determine the feasibility of this approach. If successful, the knowledge from this study can have an important impact on patients awaiting lung transplantation by providing a novel strategy for the use of HBV-positive organ donors, simplified through a shorter course of approved antivirals.

ELIGIBILITY:
Donor Inclusion Criteria

* Donor lung suitable for transplantation
* HBV SAg positive and/or HBV NAT+ donor

Donor Exclusion Criteria

* HIV positive
* HTLV 1/2 positive;
* Any medical issues in the donor that would normally clinically exclude the donor (e.g. history of cancer, evidence of organ dysfunction, etc).

Recipient inclusion Criteria:

* Recipients eligible and listed for lung transplant
* HBV NAT negative
* Provides written informed consent
* Has received at least 3 prior doses of Hepatitis B vaccine or anti-HBs>=10 IU/mL
* Patients with other co-morbid conditions (such as diabetes, autoimmune disease, renal dysfunction) will remain eligible provided they are otherwise medically suitable for transplantation. The exception to this will be patients with significant liver disease as outlined below.

Recipient exclusion Criteria:

* Chronic liver disease with > stage 2 fibrosis
* Participating in another interventional clinical trial
* Recipient listed for combined transplant (e.g., heart-lung, lung-liver)
* Known allergy or contraindication to any of the antiviral medications
* Hepatitis B surface antigen (HBsAg) or Hepatitis B core Ab positive pre-transplant (indicates already HBV infected).
* HIV positive
* Patients with a low level of serum IgA pre-transplant (this may be a risk factor for sensitivity reaction to HBIG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safety of transplantation using HBV positive donors reflected by negative HBV NAT at 6 months post-transplant | At 6 months post-transplant
  Participant blood samples will be taken at days 3 and 7, then weekly for the first 4 weeks, then every two weeks until 12 weeks post-transplant, then at month 6 after transplantation. Blood samples will be tested for HBV DNA via Nucleic Acid Amplification.

SECONDARY OUTCOMES:
Incidence of any HBV donor to recipient transmission | From enrollment until 2 years post-transplant
Correlation between donor viremia level, and recipient infection | From enrollment until up to 2 years post-transplant
Interval of time from transplantation to viremia development | From enrollment until 2 years post-transplant
HBV suppression rates after treatment for infected patients | From time of infection until end of treatment or up to 2 years post-transplant
Adverse reactions to antiviral therapy | From enrollment until 2 years post-transplant
Incidence of acute liver dysfunction for infected patients | From enrollment until 2 years post-transplant
In-hospital mortality | From hospital admission until date of discharge or date of death from any cause, whichever comes first, assessed up to 2 years
1-year graft and patient survival | Measured 1 year post-transplant
Organ function at 1 year (FEV1) | Measured 1 year post-transplant
Development of anti-HBV antibodies (anti-HBs, anti-HBc) | From enrollment until 2 years post-transplant

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No